CLINICAL TRIAL: NCT03966443
Title: PET i Diagnostikk og Behandlingsrespons av Pasienter Med Myelomatose
Brief Title: Fluciclovine PET/CT in Multiple Myeloma Patients
Acronym: FLUCIPET
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mona-Elisabeth Revheim, PI, MD, PhD, MHA, Oslo University Hospital
Other Study IDs: 2018/2212/REK
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Myeloma, Multiple; PET-CT
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparison between image findings at aminoacid PET/CT and FDG PET/CT for myeloma patients

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patients suitable for ASCT treatment

Exclusion Criteria:

* Patients with contraindications to ASCT treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple myeloma patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Comparing of image findings at PET | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hosptal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No